CLINICAL TRIAL: NCT01265693
Title: The Effect of Antiviral Therapy With Pegylated Interferon-alpha for Chronic Hepatitis C and B on Auditory Disability: A Prospective Study
Brief Title: The Effect of Antiviral Therapy With Pegylated Interferon-alpha on Auditory Disability
Acronym: HLIPT2010
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eli Zuckerman, Director of Liver Unit Carmel Medical Center, Carmel Medical Center
Other Study IDs: CMC-10-0076-CTIL
Record Dates: First submitted 2010-12-01; First posted 2010-12-23 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Hearing Loss; Sudden Deafness
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to assess the effect of antiviral therapy with pegylated interferon alpha for hepatitis C and B on auditory disability as there are reports in the English literature on auditory disability caused by interferon alpha.

DETAILED DESCRIPTION:
The population to be studied: Patients with chronic hepatitis C or B treated by pegylated interferon- alpha.

Trial Design Primary end-point: to assess the rate of auditory disability induced by pegylated interferon alpha for hepatitis C virus (HCV) and hepatitisB virus (HBV).

Secondary end-point: to investigate the outcome of auditory disability induced by pegylated interferon alpha for HCV and HBV.

Type/design of trial to be conducted: Prospective, longitudinal and controlled trial.

In each participant, base line conventional auditory assessment will be performed as well as during and at the end of treatment. The results will be compared to base-line measurements.

At base line (pre treatment), all participants will undergo a thorough conventional audiological assessment including clinical assessment by an ear, nose and throat (E.N.T) specialist and pure-tone audiometry (air conduction and if necessary also bone conduction), speech reception threshold and discrimination. In case of conductive defect detection, tympanometry will be added to auditory assessment.

Pure-tone audiometry will be re-performed at week 12 of anti-viral treatment and at the end of therapy: at week 24 in genotype 2/3 patients or at week 48 or 72 in genotype 1 patients. Additional unscheduled audiometry tests will be performed at any time during the study if a participant will complain of hearing loss or tinnitus, or as follow-up assessment in patients with treatment-induced hearing loss (as scheduled by the E.N.T specialist (co-investigator).

The following audiometric parameters will be collected:

* Pure Tone Average (PTA)- (parameter which reflects the average frequencies 500, 1000 and 2000HZ) for each ear.
* Speech Reception Threshold (SRT) for each ear.
* Discrimination values for each ear
* The degree of hearing loss (decrease in threshold sensitivity) compared with base line measurements [Δ-differences in decibels (dB)]. If hearing loss will be detected within several frequencies, the average degree of decreased sensitivity will be determined
* Presence/absence of tinnitus

Trial Objectives and Purpose To assess the rate and the outcome of auditory disability induced by pegylated interferon alpha in patients with chronic viral hepatitis C and B

Hearing loss is defined as a decrease in threshold sensitivity of 15 dB or greater at one or more test frequencies in relation to the base line measurements (in order to increase the sensitivity of hearing loss detection).

"Auditory disability" exists if either hearing loss or tinnitus occurs.

Management of anti-treatment-induced hearing loss/tinnitus:

In case of detection of hearing loss as per scheduled audiometric testing or following clinical symptoms (patient's complaints) or if tinnitus occurs, the following management will be carried out:

1. Repeated pure-tone audiometry will be performed every 5 days (up to 4 tests) as in most cases, recovery of hearing loss occurs within 2 weeks. Further need for additional follow-up audiometric testing will be determined by the investigators.
2. A discussion will be performed and documented in any case of auditory disability. The severity of hearing loss and degree of functional impairment, the results of follow-up audiometric testing, the severity of liver disease and the necessity of the continuation of anti viral therapy will be discussed.

In cases with mild, non-clinically significant and non-progressive hearing loss, continuation of anti viral therapy is optional. In that case, only follow-up measurements and testing with no further intervention will be carried out.

The need for concomitant short course of corticosteroids treatment will be discussed per each case. In cases with significant and/or progressive hearing loss or severe tinnitus, cessation of anti-viral treatment will be considered.

All participants will be identified by initials and trial number in the case report form (CRF).

Selection and Withdrawal of Subjects

Inclusion criteria:

Patients with chronic hepatitis C virus infection who will receive anti viral treatment consists of PEG-IFN-alpha-2a or 2b combined with ribavirin, Patients with chronic hepatitis B who receive anti-viral treatment with PEG-IFN-alpha 2a (Pegasys) Age 18-70 who are eligible for anti viral treatment. Patients who attend and are treated in the Liver Unit of Haifa and Western Galilee District of Clalit Health Services and Carmel Medical Center will be recruited.

Patients with all HCV genotypes will be included and will be treated by the standard-of-care therapy for hepatitis C: 48 weeks for genotypes 1 or 4.

Patients and 24 weeks for genotypes 2 or 3. Virological response will be determined at week 12 of treatment. In non-responders therapy will be discontinued.

In those patients with genotype 1 and "slow virological response", 72 weeks of therapy will be considered. Included will be also patients with chronic hepatitis B receiving PEG-IFN alpha 2a for up to 48 weeks.

Study completion is anticipated at 3 years after its initiation. Subject exclusion criteria.

1. Patients with severe base line (pre anti-viral treatment) hearing loss (>70 dB hearing levels by PTA) will be excluded.
2. Refusal to participate in the study Subject withdrawal criteria: subjects who refuse to continue participation in the study.

Assessment of Safety Auditory assessment is not associated with adverse events and it is completely safe

Statistics The distributions of continuous variables will be analyzed using the Kolmogorov-Smirnov test for normality.

The measured auditory parameters (decibels) of the patients will be compared between the three measurement times using the ANOVA test for repetitive measurements or the Friedman Two-way ANOVA test, as needed (for parametric and non-parametric groups respectively), followed by the Bonferroni post hoc test for multiple comparisons.

Categorical groups will be evaluated for associations using the Chi-square test or the Fisher's exact test, as needed.

Two-tailed p values of 0.05 or less will be considered significant. The number of subjects planned to be enrolled 100 patients. Criteria for the termination of the trial. Statistical analysis will be performed only fpr participants who will complete auditory assessment before during and at the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C virus infection who will receive anti viral treatment consists of PEG-IFN-alpha-2a or 2b combined with ribavirin,
* Patients with chronic hepatitis B who receive anti-viral treatment with PEG-IFN-alpha 2a (Pegasys)
* Age 18-70 who are eligible for anti viral treatment.
* Patients who attend and are treated in the Liver Unit of Haifa and Western
* Galilee District of Clalit Health Services and Carmel Medical Center will be recruited.
* Patients with all HCV genotypes will be included and will be treated by the standard-of-care therapy for hepatitis C: 48 weeks for genotypes 1 or 4.
* Patients and 24 weeks for genotypes 2 or 3.
* Virological response will be determined at week 12 of treatment. In non-responders therapy will be discontinued.
* In those patients with genotype 1 and "'slow virological response", 72 weeks of therapy will be considered. Included will be also patients with chronic hepatitis B receiving PEG-IFN alpha 2a for up to 48 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C or B treated with pegylated interferon alpha
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03-26 (Actual)

PRIMARY OUTCOMES:
to assess the rate of auditory disability induced by pegylated interferon alpha for HCV and HBV. | Two years

SECONDARY OUTCOMES:
to investigate the outcome of auditory disability induced by pegylated interferon alpha for HCV and HBV. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Eli Zuckerman, M.D., Principal Investigator — Liver Unit, Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No